CLINICAL TRIAL: NCT05829681
Title: Individualized Neuroimaging Biomarkers for Predicting Repetitive Transcranial Magnetic Stimulation (rTMS) Response in Obsessive Compulsive Disorder (OCD)
Brief Title: Individualized Neuroimaging Biomarkers for Predicting rTMS Response in OCD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Cornell University (Other); Foundation for OCD Research (Unknown)
Responsible Party: Principal Investigator, David Spiegel, Jack, Lulu and Sam Willson Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 62822; 22-03024635 (Other: Cornell University IRB); Pro00057331 (Other: Advarra)
Record Dates: First submitted 2023-04-06; First posted 2023-04-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: rTMS; fMRI; EEG
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Medial Prefrontal Cortex (MPFC) (Experimental): Intermittent theta-burst stimulation (iTBS) of MPFC at up to 100% resting motor threshold (RMT), with lower extremity RMT established for the MPFC target.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Right Prefrontal Cortex (rPFC) (Active Comparator): Continuous theta-burst stimulation (cTBS) of rPFC at up to 110% of RMT, with upper extremity RMT established for the rPFC target.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Participants will receive a 5-day course of 10x daily rTMS, with sessions delivered hourly. Each session will deliver up to 1800 pulses of theta-burst stimulation per target.
  Other Names: rTMS; MagVenture MagPro rTMS Research System

SUMMARY:
The goal of this clinical trial is to discover brain-based subtypes of Obsessive Compulsive Disorder (OCD) and examine treatment response to two different repetitive transcranial magnetic stimulation (rTMS) targets in the brain: the medial prefrontal cortex (MPFC) and the right prefrontal cortex (rPFC).

DETAILED DESCRIPTION:
New interventions are urgently needed to treat obsessive compulsive disorder (OCD), as more than 25% of patients show no improvement with the standard of care. Repetitive transcranial magnetic stimulation (rTMS) is a promising alternative treatment, as it uses focused magnetic field pulses to stimulate specific brain areas. So far, medial and right prefrontal cortex stimulation targets have consistent evidence of efficacy in OCD. Patients often show a strong response to one target but not the other. It is not well understood why some patients respond, while others do not. So far, there are no biomarkers for predicting treatment response, identifying the optimal neuroanatomical target, or choosing between treatments.

The goal of this clinical trial is OCD subtype discovery and treatment optimization. Using MRI scans of OCD patients before and after rTMS treatment we aim to:

* Define novel network-based subtypes of OCD that can be diagnosed in individual patients and differentiated from healthy controls;
* Identify characteristic functional connectivity profiles predictive of response to MPFC-rTMS versus rPFC-rTMS;
* Identify characteristic changes in resting-state functional connectivity (RSFC) associated with symptom improvement for OCD patients undergoing MPFC- and rPFC-rTMS.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient
2. Aged 18-80
3. Either sex and all ethno-racial categories.
4. Meets DSM-5 criteria for OCD with a moderate level of severity as defined by a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 20.
5. Off antidepressants OR on a stable dose of SRI medication for at least 8 weeks prior to the study with plans to remain on this stable dose during the study.

   a. Medications that are known to increase cortical excitability (e.g., bupropion, maprotiline, tricyclic antidepressants, classical antipsychotics) or to have an inhibitory effect on brain excitability (e.g., anticonvulsants, benzodiazepines, and atypical antipsychotics), or any other medications with relative hazard for use in TMS will be allowed upon review of medications and/or motor threshold determination by TMS specialist.
6. Failed at least 1 prior trial of standard first-line OCD treatment per APA Practice Guidelines (serotonin reuptake inhibitor [SRI] or cognitive behavioral therapy with exposure and response prevention) OR had refused these treatments for individual reasons.
7. Capacity to provide informed consent.
8. Ability to tolerate clinical study procedures.
9. Successfully complete the MRI safety screening forms without any contraindications.

Exclusion Criteria:

1. Diagnosed according to the MINI as suffering from a primary psychiatric diagnosis other than OCD.
2. Evidence of psychotic symptoms on diagnostic interview.
3. Diagnosed according to the MINI as suffering from severe Personality Disorder (excluding Obsessive-Compulsive Personality Disorder) or hospitalized due to exacerbation related to borderline personality disorder.
4. Current bipolar disorder or history of any manic episodes.
5. Current active suicidality
6. Met criteria for moderate or severe Alcohol Use Disorder, Cannabis Use Disorder, or Substance Use Disorder (except nicotine and caffeine) within the past 3 months according to DSM-5 criteria.
7. Current eating disorder
8. History of seizure, having an EEG, stroke, head injury (including neurosurgery), implanted devices, frequent or severe headaches, brain related conditions (e.g., intracranial mass lesions globe injuries, hydrocephalus), illness that caused brain injury or first degree relative with seizure disorder.
9. Significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, history of cerebrovascular accident, transient ischemic attack within two years, cerebral aneurysm, dementia, Parkinson's disease, Huntington's chorea, multiple sclerosis, epilepsy.
10. Individuals with primary hoarding disorder without a DSM-5 OCD diagnosis (as determined by MINI and YBOCS checklist).
11. Planning to commence Cognitive Behavioral Therapy (that includes exposure and response prevention) during the period of the study or have begun Cognitive Behavioral Therapy within 8 weeks prior to enrollment.
12. Pregnant or nursing females (assessed via urine dipstick), or plans to conceive during the study.
13. Positive urine screen for illicit drugs (assessed via urine dipstick) [Exceptions: (1) any prescribed medication that participant is currently taking and (2) positive cocaine metabolite after consumption of coca tea].
14. History of any implanted device or psychosurgery.
15. History of any metal in the head including the eyes and ears (outside the mouth).
16. Age of OCD symptom onset > 40.
17. History of significant hearing loss.
18. Head or neck tics which interfere with TMS and/or MRI.
19. Subjects who suffered from an unstable physical, systemic and metabolic disorder such as unstabilized blood pressure or acute, unstable cardiac disease.
20. Autism spectrum disorder
21. aTBS treatment dose > 65% maximum stimulator output (MSO)
22. Any other condition deemed by the PD to interfere with the study or increase risk to the participant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2029-03-14 (Estimated)

PRIMARY OUTCOMES:
resting-state functional connectivity (rsFC) of frontostriatal networks | pre-treatment up to 1-month post-treatment
  functional magnetic resonance imaging (fMRI) measures of resting-state functional connectivity (rsFC) in the frontostriatal networks targeted by rTMS (MPFC or rPFC)

SECONDARY OUTCOMES:
OCD symptoms | pre-treatment to 1-week post-treatment
  Change in OCD symptoms (YBOCS 2, Yale-Brown Obsessive Compulsive Scale 2, score range: 0-50, higher scores indicating higher symptom levels) following treatment with rTMS

CONTACTS AND LOCATIONS:
Overall Officials: David Spiegel, MD, Study Director — Stanford University; Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The project will implement open data dissemination to ensure that the other FFOR teams and subsequently the wider research community will have ready access to the acquired data, including clinical and neuroimaging data from patients before and after treatment. To this end, all consent forms and datasharing agreements across the recruiting sites will incorporate content to enable this open data-sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified data will be available any time following publication of outcomes from this study, with no specified end date.
Access Criteria: Deidentified data will be shared with any researcher requesting access.